CLINICAL TRIAL: NCT03498131
Title: Evaluating the Potential Role of Melatonin in Subjects With Relapsing Multiple Sclerosis (MS)
Brief Title: Melatonin in Patients With Multiple Sclerosis (MS).
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Providence Health & Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017000005
Record Dates: First submitted 2018-04-06; First posted 2018-04-13 (Actual); Results first posted 2025-02-27 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Relapsing Remitting Multiple Sclerosis
Keywords: Multiple Sclerosis; MS; Melatonin; Supplement
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — Melatonin

STUDY DESIGN:
Intervention Model Description: Subjects will be randomly assigned to receive melatonin at 3 milligrams (mg) once a day or 5mg once a day. The study drug will be taken at 21:00 each day ± 2 hours.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study is blinded to patients and providers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 3 mg Melatonin (Experimental): Subjects will receive 3 mg melatonin once a day.
  Interventions: Drug: 3 mg Melatonin
- 5 mg Melatonin (Experimental): Subjects will receive 5 mg melatonin once a day.
  Interventions: Drug: 5 mg Melatonin

INTERVENTIONS:
Drug: 3 mg Melatonin — 3 mg melatonin once each day
  Arms: 3 mg Melatonin
Drug: 5 mg Melatonin — 5 mg Melatonin once each day
  Arms: 5 mg Melatonin

SUMMARY:
To date, there are no published data on the role of melatonin supplementation or the appropriate dose for patients with multiple sclerosis. Because of the potential benefits of melatonin, this pilot study will be an exploratory investigation to evaluate the effect of supplementing melatonin in subjects with multiple sclerosis who are taking an oral disease modifying therapy (DMT) for 6 months or longer. It is our intent that the results of this study will support the rationale and be a prelude to a larger trial which can focus on clinical efficacy of melatonin therapy outcomes.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the change in 24 hour urinary 6-sulfatoxymelatonin (6SMT) collected for 24 hours in two twelve hour sessions. The secondary objectives are to evaluate the change in serum morning melatonin level. In addition, quality of life (QOL) measures will be assessed including the Modified Fatigue Impact Scale (MFIS), Multiple Sclerosis Impact Scale (MSIS-29), and the Pittsburgh Sleep Quality Index (PSQI). Clinical objectives include the number of relapses during the trial and a change in the Patient Determined Disease Steps (PDDS) & Performance Scales (PS).

The pilot study is a one-year randomized, rater- and dose-blinded trial evaluating the potential role of melatonin in subjects with relapsing multiple sclerosis who have been taking a stable dose of an oral disease modifying therapy (DMT) for at least 6 months. The oral DMTs include dimethyl fumarate, fingolimod, teriflunomide, diroximel fumarate, siponimod, and ozanimod. Thirty subjects with relapsing forms of multiple sclerosis who meet all of the eligibility criteria will be enrolled at Providence Neurological Specialties in Portland, Oregon.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects with relapsing forms of MS who have been on a stable dose of dimethyl fumarate, fingolimod, teriflunomide, diroximel fumarate, siponimod, or ozanimod for 6 months or longer
* Confirmed diagnosis of Relapsing MS
* Women of childbearing potential must employ proven methods to prevent pregnancy during the course of the trial; the acceptable method will be left to the judgment of the investigator
* Not pregnant or lactating
* No evidence of significant cognitive or psychiatric disorder
* Able to understand the purpose and risks of the study
* Must be willing to sign an informed consent and follow the protocol requirements

Exclusion Criteria:

* Use of melatonin within 30 days of enrollment
* The addition of any sleep aide or change in dose within 30 days of enrollment or during the trial
* The addition or change in dose of Vitamin D within 30 days of enrollment or during the trial
* Change in DMT during the trial
* Steroid therapy within 30 days of enrollment
* Use of anticoagulation at the time of enrollment and during the trial
* The addition of an antidepressant is not allowed during the study period; if on an antidepressant at screening, the dose must be stable 30 days prior to enrollment and dose changes are prohibited during the study
* The addition or change in dose of any stimulants, including but not limited to, amantadine, armodafinil, methylphenidate, or modafinil within 30 days of enrollment or during the trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-05-09 (Actual); Primary Completion 2022-07-29 (Actual); Study Completion 2023-12-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Smoot, MD, Principal Investigator — Providence Health & Services
Locations (1):
- Providence MS Center, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Smoot K, Gervasi-Follmar T, Marginean H, Chen C, Cohan S. Impact of oral melatonin supplementation on urine and serum melatonin concentrations and quality-of-life measures in persons with relapsing multiple sclerosis. Mult Scler Relat Disord. 2024 Oct;90:105799. doi: 10.1016/j.msard.2024.105799. Epub 2024 Aug 3. PMID 39126937
- [Derived] Ghareghani M, Farhadi Z, Rivest S, Zibara K. PDK4 Inhibition Ameliorates Melatonin Therapy by Modulating Cerebral Metabolism and Remyelination in an EAE Demyelinating Mouse Model of Multiple Sclerosis. Front Immunol. 2022 Mar 9;13:862316. doi: 10.3389/fimmu.2022.862316. eCollection 2022. PMID 35355991
- See also: Providence Brain and Spine Institute — https://oregon.providence.org/our-services/p/providence-brain-and-spine-institute/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 3 mg Melatonin | 5 mg Melatonin
Started | 15 | 15
Completed | 13 | 10
Not Completed | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 3 mg Melatonin | 5 mg Melatonin | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 57 [46 to 60] | 53 [48 to 57] | 54 [46 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 23
  Male | 3 | 4 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 15 | 15 | 30
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 15 | 14 | 29
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 15 | 30
Prior MS treatment Received [Count of Participants; unit: Participants] | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Urine Melatonin Levels
Description: Changes in urinary 6-SMT in 24 hours, urine measured in nanograms per gram of creatinine
Time Frame: Baseline (month 0), Month 3, Month 6, and Month 12
Population: Number analyzed in one or more rows differs from overall number analyzed due to patients withdrawing or being withdrawn throughout the course of the study. Numbers analyzed in serum and urine outcomes may differ in the numbers analyzed in the questionnaire outcomes (PSQI,MFIS,MSIS-29, PDDS-PS) due to patients completing questionnaires but samples not being collected or analyzed.
Measure: Median (Inter-Quartile Range); unit: nanograms per gram of creatinine
Arm/Group | 3 mg Melatonin | 5 mg Melatonin
Number analyzed (Participants) | 15 | 15
nanograms per gram of creatinine
  Baseline (month 0) | 19 [10 to 55] | 22 [16 to 91]
  Month 3: number analyzed (Participants) | 13 | 11
  Month 3 | 925 [214 to 1305] | 1,687 [808 to 4,817]
  Month 6: number analyzed (Participants) | 13 | 10
  Month 6 | 1,030 [424 to 2,245] | 2,509 [1,780 to 4,784]
  Month 12: number analyzed (Participants) | 13 | 9
  Month 12 | 1,020 [31 to 1,604] | 4,339 [653 to 16,194]

2. Secondary Outcome: Modified Fatigue Impact Scale (MFIS)
Description: Changes in the MFIS: Modified Fatigue Impact Scale (MFIS) is a PRO, consisting of 21 statements that describe the effect of fatigue. Subject will choose an answer (0= never to 4=always) that best describes how fatigue has affected them in the past 4 weeks. Item scores are summed to a total score. The total MFIS score ranges from 0 to 84, with three subscales: Physical range 0-36, Cognitive range 0-40, and Psychosocial range 0-8. Higher scores indicate higher level of fatigue.
Time Frame: Baseline (month 0), Month 3, Month 6, and Month 12
Population: Number analyzed in one or more rows differs from overall number analyzed due to patients withdrawing or being withdrawn throughout the course of the study.
Measure: Mean (Inter-Quartile Range); unit: scores on a MFIS scale
Arm/Group | 3 mg Melatonin | 5 mg Melatonin
Number analyzed (Participants) | 15 | 15
scores on a MFIS scale
  MFIS Score [0-84] - Baseline | 25 [16.0 to 25.0] | 24 [8.0 to 24.0]
  MFIS Score [0-84] - 3 months visit: number analyzed (Participants) | 14 | 11
  MFIS Score [0-84] - 3 months visit | 16.5 [9.50 to 16.5] | 22.0 [14.5 to 22.0]
  MFIS Score [0-84] - 6 months visit: number analyzed (Participants) | 14 | 10
  MFIS Score [0-84] - 6 months visit | 22 [4.75 to 22.0] | 21.5 [11.2 to 21.5]
  MFIS Score [0-84] - 12 months visit: number analyzed (Participants) | 14 | 9
  MFIS Score [0-84] - 12 months visit | 20.5 [6.00 to 20.5] | 19.0 [12.0 to 19.0]

3. Secondary Outcome: Serum Melatonin Level
Description: Changes in morning blood levels of melatonin
Time Frame: Baseline (month 0), Month 3, Month 6, and Month 12
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | 3 mg Melatonin | 5 mg Melatonin
Number analyzed (Participants) | 15 | 15
pg/ml
  Baseline (Month 0) | 5 [4 to 9] | 5 [4 to 13]
  Month 3: number analyzed (Participants) | 13 | 11
  Month 3 | 14 [8 to 44] | 69 [32 to 111]
  Month 6: number analyzed (Participants) | 13 | 10
  Month 6 | 35 [12 to 51] | 72 [46 to 193]
  Month 12: number analyzed (Participants) | 13 | 9
  Month 12 | 29 [8 to 56] | 97 [20 to 261]

4. Secondary Outcome: Multiple Sclerosis Impact Scale-29 (MSIS-29)
Description: Multiple Sclerosis Impact Scale (MSIS) is a patient reported outcome (PRO) measure, consisting of two subscales- physical impact of MS (20 items) and psychological impact (9 items). It asks subject to rate the impact MS has their daily life in the past 2 weeks (1=low impact to 4=large impact). Individual item scores are summed to create a raw score, which is then transformed on a scale from 0 to 100 for each subscale. Higher scores indicate greater impact of MS on QoL.
Time Frame: Baseline (month 0), Month 3, Month 6, and Month 12
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: MSIS-29 Score
Arm/Group | 3 mg Melatonin | 5 mg Melatonin
Number analyzed (Participants) | 15 | 15
MSIS-29 Score
  Physical - Baseline | 10 [3.00 to 10.0] | 9.00 [5.00 to 9.00]
  Physical - 3 Months Visit: number analyzed (Participants) | 14 | 11
  Physical - 3 Months Visit | 4.5 [4.00 to 4.50] | 8.00 [4.00 to 8.00]
  Physical - 6 months visit: number analyzed (Participants) | 14 | 10
  Physical - 6 months visit | 7.0 [2.50 to 7.0] | 5.00 [2.00 to 5.00]
  Physical - 12 months visit: number analyzed (Participants) | 14 | 9
  Physical - 12 months visit | 9.00 [2.00 to 9.00] | 8.00 [2.00 to 8.00]
  Psychological - Baseline | 8.0 [4.50 to 8.00] | 14.0 [9.50 to 14.0]
  Psychological - 3 months visit: number analyzed (Participants) | 14 | 11
  Psychological - 3 months visit | 12.5 [6.50 to 12.5] | 8.0 [3.00 to 8.00]
  Psychological - 6 months visit: number analyzed (Participants) | 14 | 10
  Psychological - 6 months visit | 3.0 [3.00 to 3.00] | 9.50 [8.00 to 9.50]
  Psychological - 12 months visit: number analyzed (Participants) | 14 | 9
  Psychological - 12 months visit | 8.0 [0.750 to 8.00] | 11.0 [6.00 to 11.0]

5. Secondary Outcome: Pittsburgh Sleep Quality Index (PSQI)
Description: Changes in PSQI: Pittsburgh Sleep Quality Index (PSQI) asks 10 sets of questions about sleep quality and pattern in the past month. The scale derive 7 component scores based on a 0 to 3 scale (0= no difficulty, 3=severe difficulty) which are summed to a global score (range 0 to 21). Higher scores indicates worse sleep quality.
Time Frame: Baseline (month 0), Month 3, Month 6, and Month 12
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: PSQI Score
Arm/Group | 3 mg Melatonin | 5 mg Melatonin
Number analyzed (Participants) | 15 | 15
PSQI Score
  PSQI Global - Base Line | 7.0 [5.5 to 7.0] | 6.0 [4.5 to 6.0]
  PSQI Global - 3 month Visit: number analyzed (Participants) | 14 | 11
  PSQI Global - 3 month Visit | 5.5 [3.0 to 5.5] | 9.0 [6.0 to 9.0]
  PSQI Global - 6 months visit: number analyzed (Participants) | 14 | 10
  PSQI Global - 6 months visit | 6.0 [4.0 to 6.0] | 8.0 [4.5 to 8.0]
  PSQI Global - 12 month Visit: number analyzed (Participants) | 14 | 9
  PSQI Global - 12 month Visit | 5.0 [2.5 to 5.0] | 7.0 [5.0 to 7.0]

6. Secondary Outcome: Relapse Rate
Description: Number of MS relapses during study
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | 3 mg Melatonin | 5 mg Melatonin
Number analyzed (Participants) | 15 | 15
Participants
  o Relapse | 13 | 15
  1 Relapse | 2 | 0

7. Secondary Outcome: Patient Determined Disease Steps - Performance Scale (PDDS-PS)
Description: Changes in PDDS-PS: Patient Determined Disease Steps and Performance Scales (PDDS-PS) is a PRO for MS disease status. Performance Scales (PS) has 8 subscales: mobility range, hand function range, vision range, fatigue range, cognition range, bowel/bladder range, sensory range, and spasticity range. Subject self-classify their level of disability on a 0 to 8 scale (0=Normal to 8=Bedridden) with 8 being the most disabled for PDDS. For Performance Scales (PS) subject self-classify their level of disability on a 0 to 6 scale (0=Normal to 6=Bedridden) with 6 being the most disabled for PS - Mobility. Subject self-classify their level of disability on 0 to 5 scale (0=Normal to 5=Total Disability) with 5 being the most disabled for PS - hand function range, vision range, fatigue range, cognition range, bowel/bladder range, sensory range, and spasticity range.
Time Frame: Baseline (month 0), Month 3, Month 6, and Month 12
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: scores on a PDDS-PS scale
Arm/Group | 3 mg Melatonin | 5 mg Melatonin
Number analyzed (Participants) | 15 | 15
scores on a PDDS-PS scale
  Patient Determined Disease Steps - Baseline | 1.0 [0 to 1.0] | 0 [0 to 0]
  Patient Determined Disease Steps - 3 Month Visit: number analyzed (Participants) | 14 | 11
  Patient Determined Disease Steps - 3 Month Visit | 1.0 [0 to 1.0] | 0 [0 to 0]
  Patient Determined Disease Steps - 6 Month Visit: number analyzed (Participants) | 14 | 10
  Patient Determined Disease Steps - 6 Month Visit | 0.50 [0 to 0.50] | 0.50 [0 to 0.50]
  Patient Determined Disease Steps - 12 Month Visit: number analyzed (Participants) | 14 | 9
  Patient Determined Disease Steps - 12 Month Visit | 0.50 [0 to 0.50] | 1.0 [0 to 1.0]
  Performance Scale - Mobility - Baseline | 0 [0 to 0] | 0 [0 to 0]
  Performance Scale - Mobility - 3 Month: number analyzed (Participants) | 14 | 11
  Performance Scale - Mobility - 3 Month | 0 [0 to 0] | 0 [0 to 0]
  Performance Scale - Mobility - 6 Month: number analyzed (Participants) | 14 | 10
  Performance Scale - Mobility - 6 Month | 0.500 [0 to 0.500] | 0 [0 to 0]
  Performance Scale - Mobility - 12 Month: number analyzed (Participants) | 14 | 9
  Performance Scale - Mobility - 12 Month | 0 [0 to 0] | 0 [0 to 0]
  Performance Scale - Hand Function - Baseline | 1.00 [0 to 1.00] | 0 [0 to 0]
  Performance Scale - Hand Function - 3 Month: number analyzed (Participants) | 14 | 11
  Performance Scale - Hand Function - 3 Month | 1.00 [0 to 1.00] | 0 [0 to 0]
  Performance Scale - Hand Function - 6 Month: number analyzed (Participants) | 14 | 10
  Performance Scale - Hand Function - 6 Month | 0.500 [0 to 0.500] | 0 [0 to 0]
  Performance Scale - Hand Function - 12 Month: number analyzed (Participants) | 14 | 9
  Performance Scale - Hand Function - 12 Month | 0.500 [0 to 0.500] | 0 [0 to 0]
  Performance Scale - Vision Range - Baseline | 1.00 [0 to 1.00] | 0 [0 to 0]
  Performance Scale - Vision Range - 3 Month: number analyzed (Participants) | 14 | 11
  Performance Scale - Vision Range - 3 Month | 1.00 [0 to 1.00] | 0 [0 to 0]
  Performance Scale - Vision Range - 6 Month: number analyzed (Participants) | 14 | 10
  Performance Scale - Vision Range - 6 Month | 1.00 [0 to 1.00] | 0 [0 to 0]
  Performance Scale - Vision Range - 12 Month: number analyzed (Participants) | 14 | 9
  Performance Scale - Vision Range - 12 Month | 1.00 [0 to 1.00] | 0 [0 to 0]
  Performance Scale - Fatigue - Baseline | 2.00 [1.00 to 2.00] | 2.00 [1.00 to 2.00]
  Performance Scale - Fatigue - 3 Month: number analyzed (Participants) | 14 | 11
  Performance Scale - Fatigue - 3 Month | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Performance Scale - Fatigue - 6 Month: number analyzed (Participants) | 14 | 10
  Performance Scale - Fatigue - 6 Month | 1.00 [1.00 to 1.00] | 2.00 [1.00 to 2.00]
  Performance Scale - Fatigue - 12 Month: number analyzed (Participants) | 14 | 9
  Performance Scale - Fatigue - 12 Month | 1.50 [1.00 to 1.50] | 1.00 [0 to 1.00]
  Performance Scale - Cognition Range - Baseline | 1.00 [1.00 to 1.00] | 0 [0 to 0]
  Performance Scale - Cognition Range - 3 Month: number analyzed (Participants) | 14 | 11
  Performance Scale - Cognition Range - 3 Month | 1.00 [0 to 1.00] | 0 [0 to 0]
  Performance Scale - Cognition Range - 6 Month: number analyzed (Participants) | 14 | 10
  Performance Scale - Cognition Range - 6 Month | 0.500 [0 to 0.500] | 0.500 [0 to 0.500]
  Performance Scale - Cognition Range - 12 Month: number analyzed (Participants) | 14 | 9
  Performance Scale - Cognition Range - 12 Month | 1.00 [1.00 to 1.00] | 0 [0 to 0]
  Performance Scale - Bowel/Bladder Range - Baseline | 1.00 [0.500 to 1.00] | 1.00 [0 to 1.00]
  Performance Scale - Bowel/Bladder Range - 3 Month: number analyzed (Participants) | 14 | 11
  Performance Scale - Bowel/Bladder Range - 3 Month | 0.500 [0 to 0.500] | 1.00 [0 to 1.00]
  Performance Scale - Bowel/Bladder Range - 6 Month: number analyzed (Participants) | 14 | 10
  Performance Scale - Bowel/Bladder Range - 6 Month | 1.00 [0 to 1.00] | 1.00 [0 to 1.00]
  Performance Scale - Bowel/Bladder Range - 12 Month: number analyzed (Participants) | 14 | 9
  Performance Scale - Bowel/Bladder Range - 12 Month | 1.00 [0.250 to 1.00] | 1.00 [0 to 1.00]
  Performance Scale - Sensory Range - Baseline | 1.00 [0.500 to 1.00] | 1.00 [0 to 1.00]
  Performance Scale - Sensory Range - 3 Month: number analyzed (Participants) | 14 | 11
  Performance Scale - Sensory Range - 3 Month | 1.00 [0 to 1.00] | 1.00 [1.00 to 1.00]
  Performance Scale - Sensory Range - 6 Month: number analyzed (Participants) | 14 | 10
  Performance Scale - Sensory Range - 6 Month | 1.00 [0 to 1.00] | 0.500 [0 to 0.500]
  Performance Scale - Sensory Range - 12 Month: number analyzed (Participants) | 14 | 9
  Performance Scale - Sensory Range - 12 Month | 1.00 [0 to 1.00] | 1.00 [0 to 1.00]
  Performance Scale - Spasticity - Baseline | 1.00 [0 to 1.00] | 0 [0 to 0]
  Performance Scale - Spasticity - 3 Month: number analyzed (Participants) | 14 | 11
  Performance Scale - Spasticity - 3 Month | 0 [0 to 0] | 1.00 [0 to 1.00]
  Performance Scale - Spasticity - 6 Month: number analyzed (Participants) | 14 | 10
  Performance Scale - Spasticity - 6 Month | 1.00 [0 to 1.00] | 1.00 [0 to 1.00]
  Performance Scale - Spasticity - 12 Month: number analyzed (Participants) | 14 | 9
  Performance Scale - Spasticity - 12 Month | 1.00 [0 to 1.00] | 1.00 [0 to 1.00]

ADVERSE EVENTS:
Time Frame: The period during which all adverse events and serious adverse events collected began after the informed consent is obtained and ended 30 days following the last administration of study treatment and IP assignments unblinded or study discontinuation/termination, whichever is earlier, up to 5 years.
Arm/Group | 3 mg Melatonin | 5 mg Melatonin
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 1/15 | 0/15
Other Adverse Events (participants affected / at risk) | 14/15 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3 mg Melatonin (N=15) | 5 mg Melatonin (N=15)
Near-syncope (Cardiac disorders) | 1 (1) | 0 (0)
Pacemaker insertion (Cardiac disorders) | 1 (1) | 0 (0)
Heart block (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3 mg Melatonin (N=15) | 5 mg Melatonin (N=15)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 5 (8) | 3 (4)
FLU LIKE SYMPTOMS AFTER 2ND SHINGRIX VACCINE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute Sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute viral syndrome with ageusia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute non-reccurrent frontal sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sleep Apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Essential hypertension (Cardiac disorders) | 1 (1) | 0 (0)
Type II diabetes (Endocrine disorders) | 1 (1) | 0 (0)
NIGHT SWEATS (Endocrine disorders) | 1 (1) | 0 (0)
Thyroid lobectomy (Endocrine disorders) | 0 (0) | 1 (1)
Thyroid/neck nodule increasing in size (Endocrine disorders) | 0 (0) | 1 (1)
Elevated liver function test (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Worsening hypercholesterolemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Cold Sore, Right Upper Lip (Infections and infestations) | 1 (1) | 0 (0)
POSITIVE JCV INDEX (Infections and infestations) | 1 (1) | 0 (0)
Shingles (Infections and infestations) | 1 (1) | 1 (1)
COVID Infection (Infections and infestations) | 1 (1) | 0 (0)
LOSS OF TONE/SORENESS, LEFT GLUTEUS MUSCLE (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
WORSENING OF LEG WEAKNESS, UPPER LEFT THIGH/QUAD, BILATERAL (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
SLIGHT DECREASE IN HAND DEXTERITY, LEFT (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
LOW BACK PINCHING SENSATION (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
BROKEN FINGER, LEFT HAND, 5TH FINGER (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
WEAKNESS, GENERALIZED (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Tenderness, left plantar surface of foot (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
DUPUYTREN'S CONTRACTURE, BILATERAL HANDS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Right foot pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain, lower extremities (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Weakness/tightness, lower extremities (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Medial left knee pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
RIGHT ANKLE TENDONITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Ankle sprain, left (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
STOMACH UPSET (Gastrointestinal disorders) | 1 (1) | 0 (0)
NAUSEA, SECONDARY TO WEAKNESS (Gastrointestinal disorders) | 0 (0) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 0 (0)
BOWEL URGENCY (Gastrointestinal disorders) | 1 (1) | 0 (0)
Adenomatous polyp, colon (Gastrointestinal disorders) | 1 (1) | 0 (0)
Exertional nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Increased Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
DRY MOUTH (Gastrointestinal disorders) | 1 (1) | 0 (0)
VISION CHANGES (Eye disorders) | 1 (1) | 0 (0)
Sore on tongue (Gastrointestinal disorders) | 1 (1) | 0 (0)
LESION,RIGHT POSTERIOR DORSAL TONGUE (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0)
Pharyngoesophageal dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
tooth abscess (Gastrointestinal disorders) | 0 (0) | 1 (1)
BILATERAL RECTUS RECESSION 9.0MM W/ADJUSTABLE SUTURE, LEFT EYE (Eye disorders) | 0 (0) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Temperature related pain, mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ear Infection (Ear and labyrinth disorders) | 1 (1) | 0 (0)
FATIGUE SECONDARY TO MELATONIN (General disorders) | 1 (1) | 1 (1)
WORSENING OF BALANCE ISSUES (General disorders) | 0 (0) | 1 (1)
CHILLS (General disorders) | 0 (0) | 1 (1)
HOT FLASHES (General disorders) | 0 (0) | 1 (1)
Intermittent balance issues (General disorders) | 1 (1) | 0 (0)
Shivering secondary to 2nd covid vaccine (General disorders) | 1 (1) | 0 (0)
Groggy in the mornings (General disorders) | 1 (1) | 0 (0)
Increased balance difficulties (General disorders) | 1 (1) | 0 (0)
Increased Weakness (General disorders) | 1 (1) | 0 (0)
Worsening increased weakness (General disorders) | 1 (1) | 0 (0)
Worsening increased balance difficulties (General disorders) | 1 (1) | 0 (0)
Increased fatigue (General disorders) | 1 (1) | 0 (0)
Worsening increased fatigue (General disorders) | 1 (1) | 0 (0)
BASAL CELL CARCINOMA, RIGHT CHEEK (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
PAIN SECONDARY TO BASAL CELL CARCINOMA REMOVAL, RIGHT CHEEK (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
BASAL CELL CARCINOMA, RIGHT CHEEK, REMOVAL (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
SENSORY DISTURBANCE RIGHT CHEEK, SECONDARY TO BASAL CELL CARCINOMA REMOVAL (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
WELL HEALED SCAR SECONDARY TO BASAL CARCINOMA REMOVAL (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
SPITZ NEVUS,RIGHT ANTERIOR LATERAL ARM, BIOPSY (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
NEOPLASM, UNSPECIFIED, BIOPSY RIGHT ANTERIOR LATERAL ARM (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
DERMATOFIBROMA, RIGHT BUTTOCK (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
LENTIGO (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
CHERRY ANGIOMA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
XEROSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
SPITZ NEVUS, RIGHT ANTERIOR LATERAL ARM (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
GIANT COMEDONE (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
SEBORRHEIC KERATOSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash, lower left buttocks (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Mild edema, bilateral legs (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Focal spongiotic dermatitis with many eosinophils (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Worsening of rash, multiple diffuse locations (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
SKIN SPLIT BETWEEN D1 AND D2 RIGHT FOOT (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
GENERALIZED DRYNESS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Contact dermatitis, nose (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Cyst removal incision infection, back (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Cyst removal, back (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Epidemal inclusion cyst (Surgical and medical procedures) | 0 (0) | 1 (1)
Onychomyosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Tinea pedis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash, facial (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Scaring, extremities (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
left labial cysts (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Toe nail fungus, right (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
General pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Chilblains, bilateral arms (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Squamous cell in situ, scalp (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
POSSIBLE URINARY TRACT INFECTION (Renal and urinary disorders) | 0 (0) | 1 (1)
POSSIBLE URINARY RETENTION (Renal and urinary disorders) | 0 (0) | 1 (1)
INTERMITTENT IRREGULAR MENSTRUAL CYCLES (Renal and urinary disorders) | 1 (1) | 0 (0)
IRREGULAR MENSTRUAL BLEEDING (Renal and urinary disorders) | 1 (1) | 0 (0)
Increased urinary urgency (Renal and urinary disorders) | 1 (1) | 1 (1)
Yeast infection (Renal and urinary disorders) | 0 (0) | 1 (1)
Cervical friability/lesion (benign) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
vaginal prolapse (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urinary tract infection (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (2)
Intermittent Urinary Hesitancy (Renal and urinary disorders) | 1 (1) | 0 (0)
WORSENING OF FATIGUE (Psychiatric disorders) | 0 (0) | 1 (1)
INCREASED FATIGUE (Psychiatric disorders) | 3 (3) | 0 (0)
IRRITABILITY (Psychiatric disorders) | 2 (2) | 0 (0)
WORSENING DEPRESSION (Psychiatric disorders) | 1 (1) | 2 (2)
RESTLESS SLEEP (Psychiatric disorders) | 0 (0) | 1 (1)
SLEEP ISSUES (Psychiatric disorders) | 1 (1) | 0 (0)
INCREASED DREAMING (Psychiatric disorders) | 1 (1) | 0 (0)
Increased stress (Psychiatric disorders) | 1 (1) | 0 (0)
Worsening insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Increased anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Intermittent sleep issues (Psychiatric disorders) | 0 (0) | 1 (1)
SLEEP DISTURBANCES (Psychiatric disorders) | 0 (0) | 1 (1)
ANXIETY/MOOD DISTURBANCES (Psychiatric disorders) | 0 (0) | 1 (1)
Restless during the night, unable to fall asleep (Psychiatric disorders) | 1 (1) | 0 (0)
TWO NEW ENHANCING BRAIN LESIONS (Nervous system disorders) | 0 (0) | 1 (1)
WORD FINDING ISSUES (Nervous system disorders) | 0 (0) | 1 (1)
RADIATING PAIN, LOW BACK DOWN RIGHT LEG (Nervous system disorders) | 0 (0) | 1 (1)
INTERMITTENT TINGLING BILATERAL FEET (Nervous system disorders) | 0 (0) | 1 (1)
CONCUSSION (Nervous system disorders) | 1 (1) | 0 (0)
DIZZINESS, SECONDARY TO WEAKNESS (Nervous system disorders) | 0 (0) | 1 (1)
Intermittent dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
INCREASED HEADACHES (Nervous system disorders) | 2 (2) | 0 (0)
INCREASED RESTLESS LEG SYNDROME (Nervous system disorders) | 1 (1) | 0 (0)
NUMBNESS BACK OF TONGUE (Nervous system disorders) | 1 (1) | 0 (0)
INTERMITTENT SENSORY DISTURBANCE, HEAD (Nervous system disorders) | 1 (1) | 0 (0)
Increased numbness, toes (Nervous system disorders) | 1 (1) | 0 (0)
Trigeminal neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
headaches upon waking in morning (Nervous system disorders) | 1 (1) | 0 (0)
Worsening Memory Disorder (Nervous system disorders) | 1 (1) | 0 (0)
Worsening Trigeminal Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Carpel tunnel, left (Nervous system disorders) | 1 (1) | 0 (0)
Median Neuropathy, Left Hand (Nervous system disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
1. Size of the patient population due to budget concerns.
2. No placebo arm, but the baseline values before the first dose of melatonin administration allowed each patient to severe as an internal control.
3. The time of year was not accounted for in analyzing the data.
4. The study was conducted during the SARS-CoV-2 pandemic leading to several missed data points.
5. A high number of patients that discontinued treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-09): https://cdn.clinicaltrials.gov/large-docs/31/NCT03498131/Prot_SAP_000.pdf